CLINICAL TRIAL: NCT05873153
Title: Reducing Cardiovascular Disparities in the Greater Mankato Somali Community by Utilizing Community-based Interventions to Build Capacity Within the Community to Identify, Manage and Prevent Hypertension
Brief Title: A Study of Cardiovascular Disparities in the Greater Mankato Somali Community to Prevent Hypertension
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Erin C. Westfall, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-003544; P50MD017342 (NIH)
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): Participants will be given access to health education, home blood pressure monitor, and referral to a primary care provider.
  Interventions: Behavioral: Health Education; Other: Home Blood Pressure Monitor
- Control Group (No Intervention): Participants receive referrals only to a primary care provider (PCP) for blood pressure monitoring.

INTERVENTIONS:
Behavioral: Health Education — Education materials on high blood pressure, lowering sodium, starting an exercise program, and weight management.
  Arms: Treatment Group
Other: Home Blood Pressure Monitor — Blood pressure cuff for home use
  Arms: Treatment Group

SUMMARY:
The purpose of this research is to develop ways to reduce hypertension-management-related disparities in the Greater Mankato Area Somali population.

DETAILED DESCRIPTION:
* We will randomly assign participants to either the treatment or control group. Participants in the treatment group will be given access to the education or BP monitor. Participants in the control group will receive referrals only to a PCP. We will use pre- and post-intervention to examine baseline data (during randomization) and assess changes in BP status and PCP follow up. A 3 weeks and 3 months assessment will determine BP control and PCP status. By comparing between pre- and post-intervention data, we can identify whether the educational content is effective in improving participants' knowledge, attitude, and health seeking behavior for high BP. By comparing between the treatment and control groups, we can examine to what extent the education and BP monitoring influences the effectiveness of the educational intervention.
* We will assess reach by tracking and recording the number of community members screened at each screening station, the Mosque and Halal Store. Each person will only be screened at baseline, 6 weeks and 3 months and we will record their systolic and diastolic blood pressures, age, sex, PCP status, and most recent visit with a healthcare provider. Additionally, the CHW will follow up with those that were referred for education and/or PCP visit to identify how many followed through with the recommendations (daily BP check, 30 minutes physical activity, dietary changes). Interviews will be conducted with community members who were referred to PCP and health educators due to high BP to assess the impact of the CHW/educators on their health seeking behaviors including motivation to make changes such as checking blood pressures, making dietary changes, increasing physical activity and seeking primary care, as well as how their experience with peer education was. CHW will also be interviewed to understand their overall perception of screening, suggestions for improvement. Following a community members referral to the champions for acute care needs (if they don't have a PCP or are unable to get in in a timely manner), participants' feedback about their visit with the provider will be collected to assess their overall experience with the provider.

Approach for Aim 2: Test the effectiveness of training Halal staff and Somali leaders to educate community members regarding culturally appropriate dietary recommendations and other lifestyle interventions for hypertension. For this aim Halal store owners and community leaders will keep a weekly record of the number of community members they reached out to. Additionally, community members who receive peer education will be interviewed to determine if the education from the Halal store owners was helpful, and what their experience was like Halal store owners and community leaders will also be interviewed to assess their overall perception of the peer education.

Approach for Aim 3: Build research capacity within the GMHEP members to engage in community-based research projects. Focus group will be conducted with GMHEP members following educational session to determine their experience with research education and comfort with conducting focus groups to peers.

ELIGIBILITY:
Inclusion Criteria:

* Greater Mankato Somali community members.
* Non-pregnant.
* At the Mosque or Halal stores between 5/2/2022-5/31/2023.

Exclusion Criteria:

* Pregnant.
* Are not at the Mosque or Halal stores between 5/2/2022-5/31/2023.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in systolic and diastolic blood pressure | Baseline, 3 weeks, 3 months
  Measured in millimeters of mercury (mmHg) of Systolic and Diastolic Blood pressure
Change in Primary Care Provider status | Baseline, 3 weeks, 3 months
  Number of subjects to follow up with a primary care provider

CONTACTS AND LOCATIONS:
Overall Officials: Erin Westfall, DO, Principal Investigator — Mayo Clinic
Locations (1):
- Erin Westfall, Mankato, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: clinical trials.gov — http://clinicaltrials.gov/